CLINICAL TRIAL: NCT04039087
Title: Mechanisms of Exercise Intolerance in Cystic Fibrosis: Role of PDE5 Inhibition
Brief Title: Sildenafil Exercise: Role of PDE5 Inhibition
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Augusta University (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Taylor-Cousar, Medical Director, Clinical Research Services; Professor, Departments of Medicine and Pediatrics,, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Sildenafil Exercise
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
Keywords: Exercise intolerance; Quality of life; Cardiac function
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to the sildenafil or placebo groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care provider, investigator and those assessing the outcomes will be blinded to treatment designation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Active Comparator): active sildenafil 40 mg p.o. three times per day
  Interventions: Drug: Sildenafil 40mg oral capsule
- Placebo Arm (Placebo Comparator): placebo three times per day
  Interventions: Drug: Placebo Oral capsule

INTERVENTIONS:
Drug: Sildenafil 40mg oral capsule — 40 mg, sildenafil capsule taken by mouth thrice daily
  Other Names: sildenafil, revatio
  Arms: Sildenafil
Drug: Placebo Oral capsule — Placebo capsule taken by mouth thrice daily
  Other Names: placebo
  Arms: Placebo Arm

SUMMARY:
Exercise intolerance is an understudied phenomenon in people with CF. The investigators hypothesized that vascular dysfunction plays a significant role, and can be partially reversed by administration of the phosphodiesterase type 5 (PDE5) inhibitor, sildenafil.

DETAILED DESCRIPTION:
While cystic fibrosis (CF) is most common in people of European ancestry, it can occur in individuals of any ethnicity. The predicted median life expectancy age for patients with CF is 47.7 years compared to 78.8 years in the general U.S. population. Exercise intolerance, evaluated as a reduction in exercise capacity (VO2 peak), has been shown to predict mortality in patients with CF independent of lung function. A critical barrier to improving exercise tolerance in CF is the lack of knowledge regarding the different physiological mechanisms which contribute to decreased exercise capacity. The present investigation will not only evaluate the impact that sildenafil has on clinically relevant and patient oriented outcomes, it will also provide mechanistic insight.

Phosphodiesterase type 5 (PDE5) inhibitors reduce inflammation, improve vascular health, increase microvascular O2 delivery and improve skeletal muscle function. Accordingly, the central hypothesis of the study is that treatment with the PDE5 inhibitor, sildenafil, can improve exercise capacity, vascular and cardiac function, and overall quality of life, all of which may contribute to improvement in exercise tolerance in people with CF

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis (CF) based on the following criteria: Positive sweat chloride concentration ≥60 milliequivalents (mEq)/liter (by pilocarpine iontophoresis) and/or genotype with two identifiable disease-causing mutations consistent with CF, and accompanied by one or more clinical features consistent with the CF phenotype
* Male or female patients ≥ 9 years of age
* forced expiratory volume at one second (FEV1) ≥ 30% predicted and ≤ 70% for patients ≥ 18 years of age and ≤ 80% for patients ≥ 18 years of age
* Clinically stable without evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the 14 days prior to the screening visit
* Resting oxygen saturation (room air) >85%
* Patients with or without CF related diabetes
* Ability to perform spirometry reproducibly (according to American Thoracic Society criteria)
* Willingness to maintain chronic CF medication schedule (e.g. alternating month inhaled antibiotics)

Exclusion Criteria:

* Children 8 yrs. old and younger
* Subjects who weigh < 20 Kgs
* History of hypersensitivity to sildenafil
* Use of an investigational agent within the 4-week period prior to Visit 1 (Day 0)
* Breastfeeding, pregnant, or verbal expression of unwillingness to practice an acceptable birth control method (abstinence, hormonal or barrier methods, partner sterilization or intrauterine device) during participation in the study for women of child-bearing potential.
* History of significant hepatic disease (aspartate transaminase or alanine transaminase > 3 times the upper limit of normal at screening, documented biliary cirrhosis, or portal hypertension),
* History of significant cardiovascular disease (history of aortic stenosis, coronary artery disease, or life-threatening arrhythmia),
* History of severe neurological disease (e.g. history of stroke),
* History of severe hematologic disease (e.g. history of bleeding diathesis; current international normalized ratio (INR) > 2.0
* History of severe ophthalmologic disease (e.g. history of retinal impairment or non-arteritic ischemic optic neuritis)
* History of severe renal impairment (creatinine >1.8 mg/dL.)
* Inability to swallow pills
* Previous organ transplantation
* Use of concomitant nitrates, α-blocker, or Ca channel blocker (currently or within one month of Visit 1)
* Use of concomitant medications known to be potent inhibitors of CYP3A4 [e.g. ketoconazole, itraconazole, ritonavir, clarithromycin, erythromycin, rifampin (currently or within one month of initiation of study drug)] (NOTE: use of azithromycin is NOT a cause for exclusion)
* History of sputum or throat swab culture yielding Burkholderia cepacia or Mycobacteria massiliense within 2 years of screening
* History of migraine headaches.
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data
* Initiation of a cystic fibrosis transmembrane conductance regulator (CFTR) modulator therapy less than 1 month prior to first dose of sildenafil or placebo
* Use of anticoagulants
* Frank pulmonary hypertension[right ventricular systolic pressure (RVSP) >40 mm Hg by echocardiography)
* History of Priapism or known penile anatomical deformities

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Distance (6MWD) | Change in distance walked between week 1 and week 12.
  capacity, an objective measurement of exercise tolerance, predicts mortality in patients with CF. The mechanisms for exercise intolerance in CF have yet to be fully elucidated and further understanding could improve clinical outcomes and survival in CF. Preliminary data from two independent proof-of-concept clinical trials support the use of sildenafil to improve exercise capacity, cardiac function, and quality of life in CF

SECONDARY OUTCOMES:
Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory domain score | Quality of life assessed at weeks 1 and 12.
  The respiratory domain of the validated CF-specific quality of life measure. The CFQ-R Respiratory domain score (scale 0-100 with higher scores indicating better quality of life).
Cardiac strain | Change in cardiac strain between weeks 1 and 12
  Right ventricular strain will be calculated from cardiac magnetic resonance image (MRI)
Flow-Mediated Dilation (FMD) | Change in FMD between weeks 1 and 12
  Brachial artery FMD induced by reactive hyperemia will be used to assess vascular endothelial function.
Skeletal muscle function | Change in skeletal muscle function between weeks 1 and 12
  Near infrared spectroscopy (NIRS) placed over the vastus lateralus and gastrocnemius will be used to measure changes in skeletal muscle O2 concentrations and consumption at rest and during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Taylor-Cousar, MD, MSCS, Principal Investigator — National Jewish Health
Locations (2):
- United States (2):
  - National Jewish Health, Denver, Colorado
  - Augusta University, Augusta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor-Cousar JL, Wiley C, Felton LA, St Clair C, Jones M, Curran-Everett D, Poch K, Nichols DP, Solomon GM, Saavedra MT, Accurso FJ, Nick JA. Pharmacokinetics and tolerability of oral sildenafil in adults with cystic fibrosis lung disease. J Cyst Fibros. 2015 Mar;14(2):228-36. doi: 10.1016/j.jcf.2014.10.006. Epub 2014 Nov 13. PMID 25466700
- [Background] Rodriguez-Miguelez P, Lee N, Tucker MA, Csanyi G, McKie KT, Forseen C, Harris RA. Sildenafil improves vascular endothelial function in patients with cystic fibrosis. Am J Physiol Heart Circ Physiol. 2018 Nov 1;315(5):H1486-H1494. doi: 10.1152/ajpheart.00301.2018. Epub 2018 Aug 31. PMID 30168731